CLINICAL TRIAL: NCT01641861
Title: Study of Papacarie® for Caries Removal.
Brief Title: A Comparative Study of Papacarie® and the Conventional Method for Dental Caries Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Kemporn Kitsahawong, Associated Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE542161; D43TW007768 (NIH)
Record Dates: First submitted 2012-07-09; First posted 2012-07-17 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2015-12

CONDITIONS: Dental Caries; Secondary Dental Caries; Personal Satisfaction
Keywords: Chemo-mechanical caries removal; Papacarie®
MeSH Terms: conditions — Dental Caries; Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Experimental): control arm is dental caries removal using the conventional method. Dental caries will be removed using rotary instrument following the usual procedures employed by the dentist.
  Interventions: Procedure: Conventional method
- Intervention arm (Experimental): Intervention arm is dental caries removal using Papacarie®. The dentist will apply Papacarie® to dental cavity in order to soften the carious dentine. Dental caries will be removed using hand instrument.
  Interventions: Device: Papacarie®

INTERVENTIONS:
Device: Papacarie® — Papacarie® is chemo-mechanical method for caries removal
  Other Names: Chemo-mechanical removal of decays Agent
  Arms: Intervention arm
Procedure: Conventional method — caries removal by using rotary instrument.
  Arms: Control arm

SUMMARY:
The purpose study are to evaluate the efficacy of Papacarie® for caries removal in comparison to the conventional drilling method.

DETAILED DESCRIPTION:
Dental caries in children continues to affect a significant portion of the world population, especially in developing countries. There are many techniques used for dental caries treatment. The conventional method is to remove caries and prepare the cavity using dental burs. Disadvantages of this method; however, include the patients' repulsion of drilling, and possible thermal changes on tooth surface that may have an effect on the dental pulp tissues. In addition, the drilling technique frequently requires local anesthesia injections and sometimes results in the removal of sound tooth tissues. To overcome these problems and preserve the healthy dental tissues, the chemo-mechanical caries removal method was developed. The advantage by chemomechanical caries removal include less traumatic, less need local anesthesia, reduced chance of dental pulp exposure. And also it could be benefit to medical compromised patients.

Papacarie® is a new chemo-mechanical technique for caries removal with few published research and case reports. A randomized controlled trial is therefore needed to determine the efficacy of its use in general population. The aims of this study are to evaluate the efficacy of a chemo-mechanical system (Papacarie®) for caries removal in comparison to the conventional drilling method.

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion criteria:
* Child is between 7-8 years of ages (at date of enrollment) with at least one active caries lesion in second primary molar tooth with distinct dentine involvement requiring restoration
* Child is in good general health and has no existing health condition that may interfere with treatment such as asthma, tuberculosis, rheumatic fever/ congenital heart diseases, jaundice, juvenile diabetes, haemophilia, thalassemia, leukemia, anemia , HIV , allergy to any drug, and epilepsy.
* Tooth inclusion criteria:
* Second primary molar tooth with one active caries lesion with distinct dentine involvement requiring restoration using the World Health Organization Criteria.
* Tooth with isolated occlusal caries and caries extended on further than two-third of the dentine layer, which can be restoration as a Class I restoration.
* Carious cavity must be large enough so that the hand instruments can be operated.
* Tooth is vital without pathological process assessed clinically and radiographically.

Exclusion Criteria:

* Patient exclusion criteria:
* Child whose parent does not give informed consent.
* Child who are unwilling to undergo the dental treatment.
* Child who has a known allergy to the ingredients contained in dental anesthesia, Papacarie® or glass-ionomer filling material.
* Tooth exclusion criteria:
* Having extensive dental caries which may require pulp treatment.
* Tooth with a pathological process of the dental tissue other than caries that could affect the treatment, such as tooth development disorders or adjacent soft tissue lesion.

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 488 (Actual)
Dates: Start 2012-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kemporn Kitsahawong, DDS., MSc., Principal Investigator — Faculty of Dentistry, Khon Kaen University
Locations (1):
- Faculty of Dentistry , Khon Kaen University, Muang, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kitsahawong K, Seminario AL, Pungchanchaikul P, Rattanacharoenthum A, Sutthiprapaporn P, Pitiphat W. Efficacy of chemo-mechanical caries removal: a 24-month randomized trial. Front Oral Health. 2024 Dec 3;5:1458530. doi: 10.3389/froh.2024.1458530. eCollection 2024. PMID 39697785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consists of students attending primary schools in Khon Kaen province, Thailand. Consented children were obtain clinical and radiographic examination at the Pediatric Department, Faculty of Dentistry, Khon Kaen University (KKU) in order to evaluate for their eligibility. The recruitment period were November 2012 to August 2013.
Pre-assignment Details: Among of 1299 children provided the consent and received an oral examination, 518 children received a radiographic examination for definite diagnosis. From 494 eligible children, 488 have been enrolled. The rest were not enrolled either because of parental refusal (n=2), child refusal (n=3), or the child moved to another province (n=1).
Period: Overall Study
Arm/Group | Control Arm | Intervention Arm
Started | 246 | 242
Completed | 211 | 217
Not Completed | 35 | 25
Not completed — Lost to Follow-up | 21 | 16
Not completed — Lost the tooth due to normal exfoliation | 14 | 8
Not completed — Died due to drowning | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention Arm | Total
Number analyzed (Participants) | 246 | 242 | 488
Age, Continuous [Mean (Standard Deviation); unit: months] | 89.9 (8.4) | 89.2 (7.5) | 89.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 116 | 245
  Male | 117 | 126 | 243

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Failure
Description: The dental restorations were evaluated at 6, 12, 18 and 24 months after treatment. Evaluation criteria included the condition of the filling material and presence of secondary caries at the margin of the restorations. The restoration status was re-categorized as a binary outcome: Treatment failure (Yes/No).
Time Frame: two years
Measure: Number; unit: participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 211 | 217
participants | 2 | 2
Statistical Analysis 1: Comparison: Control Arm vs Intervention Arm; Test type: Superiority or Other; Odds Ratio (OR) = 1, 95% CI 2-sided [0.1 to 7.3]

2. Secondary Outcome: Incidence of Secondary Caries
Description: The restoration teeth were assess by clinical and radiographic examination for detection the recurrent caries.
Time Frame: two years
Measure: Number; unit: participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 211 | 217
participants | 3 | 10
Statistical Analysis 1: Comparison: Control Arm vs Intervention Arm; Test type: Superiority or Other; Odds Ratio (OR) = 3.5, 95% CI 2-sided [0.9 to 12.8]

3. Secondary Outcome: Number of Participants With Complete Caries Removal
Description: The efficacy of caries removal was evaluated by the visual and tactile criteria. The completeness of caries removal was judged on the basis of clinical criteria involving the inspection of the tooth surfaces using a good light source, dental mirror and explorer. A blunt explorer was used to detect surface roughness by gently stroking across the dentine surfaces and to evaluate the dentine hardness. Complete caries removal was achieved if as remove soft and infected dentine until felt hard and leathery consistency of the dentine surfaces. The tactile criteria include the smooth passage of the blunt explorer and absence of a catch or a "tug-back" sensation.
Time Frame: immediately after treatment
Measure: Number; unit: participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 246 | 242
participants | 246 | 242

4. Secondary Outcome: Levels of Pain and Discomfort
Description: The participants were assessed for the levels of pain and discomfort using the facial visual analogue scale (VAS). The score was recorded in ruler scale from 0-100 millimeters, 0 = no pain and 100 = extreme pain) before treatment with the child sitting on the dental chair and after treatment (completion of carious tissue removal). The difference in the VAS scores before and after treatment was calculated and compared between the two comparison groups.
Time Frame: immediately after treatment
Measure: Median (Inter-Quartile Range); unit: Pain score from 0-100
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 246 | 242
Pain score from 0-100 | 25 [17 to 37] | 10 [0 to 18]
Statistical Analysis 1: Comparison: Control Arm vs Intervention Arm; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Time Use for Caries Removal
Description: The time taken for the removal of carious dentine was recorded using a stopwatch. Recorded time unit is seconds.
Time Frame: Immediately while treatment
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 246 | 242
seconds | 103 [92 to 152] | 512 [404 to 637]
Statistical Analysis 1: Comparison: Control Arm vs Intervention Arm; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at follow up visit every six months until two years.
Arm/Group | Control Arm | Intervention Arm
Serious Adverse Events (participants affected / at risk) | 0/246 | 0/242
Other Adverse Events (participants affected / at risk) | 0/246 | 0/242

LIMITATIONS AND CAVEATS:
The limitations: First, the long duration of the trial caused participants to lost to follow up. Second, the operator and patients could not be blinded from the treatment status because of the apparent difference in the intervention techniques.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No